CLINICAL TRIAL: NCT04951063
Title: Fraction Dose Escalation of Hypofractionated Radiotherapy With Concurrent Chemotherapy and Subsequent Consolidation Immunotherapy in Locally Advanced Non-small Cell Lung Cancer: a Phase 1 Study
Brief Title: Fraction Dose Escalation of Hypo-fractionated Radiotherapy in LANSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1080
Record Dates: First submitted 2021-06-26; First posted 2021-07-06 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced Lung Carcinoma
Keywords: Locally advanced non-small cell lung cancer; Definitive hypofractionated chemoradiotherapy; Fraction dose escalation; Consolidation immunotherapy
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Split-course adaptive HRT-CHT (Experimental): In keeping the same total radiation dose (60Gy), we escalate the fraction dose to find the maximum tolerable fraction dose.
  1. Level 1: DT 4500cGy/15 daily fractions/300cGy in the first course，DT 1500cGy/5 daily fractions/300cGy in the second course;
  2. Level 2: DT 4000cGy/10 daily fractions/400cGy in the first course， DT 2000cGy/5 daily fractions/400cGy in the second course;
  3. Level 3: DT 3000cGy/6 daily fractions/500cGy in the first course， DT 3000cGy/6 daily fractions/500cGy in the second course.
  RT is delivered using the IMRT technique with daily cone-beam CT image guidance. The dose limitation of organ at risk (OAR) are shown in Table 1. Patients receive a weekly infusion of docetaxel (25mg/m2) and cisplatin (25mg/m2) during RT. Consolidative immunotherapy (PD-1 or PD-L1 inhibitor) up to 1 year is administered for those without disease progression after HRT-CHT.
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: Concurrent chemotherapy; Drug: Consolidation immunotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Split-course adaptive HRT-CHT is administered at the following three dose levels:
  1. Level 1: DT 4500cGy/15 daily fractions/300cGy in the first course，DT 1500cGy/5 daily fractions/300cGy in the second course;
  2. Level 2: DT 4000cGy/10 daily fractions/400cGy in the first course， DT 2000cGy/5 daily fractions/400cGy in the second course;
  3. Level 3: DT 3000cGy/6 daily fractions/500cGy in the first course， DT 3000cGy/6 daily fractions/500cGy in the second course.
Drug: Concurrent chemotherapy — weekly infusion of docetaxel (25mg/m2) and cisplatin (25mg/m2) during RT
Drug: Consolidation immunotherapy — Consolidative immunotherapy (PD-1 or PD-L1 inhibitor) up to 1 year is administered for those without disease progression after HRT-CHT.

SUMMARY:
This Phase 1 trial aimed to determine the maximum tolerated fraction dose (MTD) of hypofractionated radiotherapy (hypo-RT) combined with concurrent chemotherapy and subsequent consolidation immune checkpoint inhibitors (cICI) for patients with locally advanced non-small cell lung cancer (LA-NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer confirmed by histology.
* Tumor size is measured according to RECIST standard.
* Unresectable stage IIIA (N2) and IIIB/IIIC, confirmed by PET-CT/or chest and abdomen CT, brain MRI, and whole body bone scan.
* 18-75 years old, regardless of gender.
* The ECOG score is 0-1.
* Newly treated or underwent neoadjuvant chemotherapy and/or immunotherapy.
* Have not received chest radiotherapy in the past.
* Serum hemoglobin ≥10 mg/dL, platelets ≥100000/μL, absolute neutrophil count ≥1500/μL.
* Serum creatinine ≤1.25 times UNL or creatinine clearance ≥60 ml/min.
* Serum bilirubin ≤1.5 times UNL, AST (SGOT) and ALT (SGPT) ≤2.5 times UNL, alkaline phosphatase≤ 5 times UNL.
* FEV1>1 L.
* CB6 normal range.
* The patient and his family members agree and sign an informed consent form.

Exclusion Criteria:

* Other malignant tumors in the past or during treatment, except for non-melanoma of the skin or carcinoma in situ of the cervix.
* Any other diseases or conditions are contraindications to chemotherapy (such as active infection, within 6 months after myocardial infarction, symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia, immunosuppressive therapy).
* Pregnant or breastfeeding women, women who have not undergone a pregnancy test (within 14 days before the first dose), and pregnant women.
* Those who are pregnant, breastfeeding or have fertility but have not taken contraceptive measures.
* People with bleeding tendency.
* Those who participated in other clinical trials within 30 days before participating in this experiment.
* Drug addiction, long-term alcoholism, and AIDS patients.
* People with uncontrollable seizures or loss of self-control due to mental illness.
* People with a history of severe allergies or specific physique.
* The researcher believes that the patient is inappropriate to participate in this trial.

Exit criteria

* The treatment cannot be carried out in accordance with the requirements of the research protocol;
* The patient has an allergic reaction ≥ grade 4 or a serious adverse reaction to the study drug;
* The patient is pregnant or has not used adequate contraceptive measures;
* The researcher judges that the patient should not continue to participate the clinical trial;
* The subject asked to withdraw.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
the maximally tolerated fraction dose | 1 year
  The maximum tolerated fraction dose was defined as the highest DL in which <=2 patients of the 6 treated patients experienced G3+ toxicity and <=1 patient experienced G4+ toxicity within 12 months after RT. If a patient had multiple types of toxicities, only the highest grade of toxicity was counted.

SECONDARY OUTCOMES:
Objective response rate | 2 months after radiotherapy
  Proportion of patients with PR and CR at 2 months after radiotherapy
Overall survival | 1-year
Progression-free survival | 1-year
Distant-metastasis free survival | 1-year
Loco-regional recurrence-free survival | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Gray JE, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, Cho BC, Planchard D, Paz-Ares L, Faivre-Finn C, Vansteenkiste JF, Spigel DR, Wadsworth C, Taboada M, Dennis PA, Ozguroglu M, Antonia SJ. Three-Year Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC-Update from PACIFIC. J Thorac Oncol. 2020 Feb;15(2):288-293. doi: 10.1016/j.jtho.2019.10.002. Epub 2019 Oct 14. PMID 31622733
- [Background] Cannon DM, Mehta MP, Adkison JB, Khuntia D, Traynor AM, Tome WA, Chappell RJ, Tolakanahalli R, Mohindra P, Bentzen SM, Cannon GM. Dose-limiting toxicity after hypofractionated dose-escalated radiotherapy in non-small-cell lung cancer. J Clin Oncol. 2013 Dec 1;31(34):4343-8. doi: 10.1200/JCO.2013.51.5353. Epub 2013 Oct 21. PMID 24145340
- [Background] Uitterhoeve AL, Belderbos JS, Koolen MG, van der Vaart PJ, Rodrigus PT, Benraadt J, Koning CC, Gonzalez Gonzalez D, Bartelink H. Toxicity of high-dose radiotherapy combined with daily cisplatin in non-small cell lung cancer: results of the EORTC 08912 phase I/II study. European Organization for Research and Treatment of Cancer. Eur J Cancer. 2000 Mar;36(5):592-600. doi: 10.1016/s0959-8049(99)00315-9. PMID 10738123
- [Background] Graham MV, Pajak TE, Herskovic AM, Emami B, Perez CA. Phase I/II study of treatment of locally advanced (T3/T4) non-oat cell lung cancer with concomitant boost radiotherapy by the Radiation Therapy Oncology Group (RTOG 83-12): long-term results. Int J Radiat Oncol Biol Phys. 1995 Feb 15;31(4):819-25. doi: 10.1016/0360-3016(94)00543-5. PMID 7860394
- [Background] Qiu B, Li QW, Ai XL, Wang B, Huan J, Zhu ZF, Yu GH, Ji M, Jiang HH, Li C, Zhang J, Chen L, Guo JY, Zhou Y, Liu H. Investigating the loco-regional control of simultaneous integrated boost intensity-modulated radiotherapy with different radiation fraction sizes for locally advanced non-small-cell lung cancer: clinical outcomes and the application of an extended LQ/TCP model. Radiat Oncol. 2020 May 27;15(1):124. doi: 10.1186/s13014-020-01555-x. PMID 32460796
- [Background] Glinski K, Socha J, Wasilewska-Tesluk E, Komosinska K, Kepka L. Accelerated hypofractionated radiotherapy with concurrent full dose chemotherapy for locally advanced non-small cell lung cancer: A phase I/II study. Radiother Oncol. 2020 Jul;148:174-180. doi: 10.1016/j.radonc.2020.04.033. Epub 2020 Apr 24. PMID 32388152
- [Background] Kong C, Zhu X, Shi M, Wang L, Chen C, Tao H, Jiang N, Yan P, Zhao L, Song X, He X. Survival and Toxicity of Hypofractionated Intensity Modulated Radiation Therapy in 4 Gy Fractions for Unresectable Stage III Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):710-719. doi: 10.1016/j.ijrobp.2020.03.038. Epub 2020 Apr 7. PMID 32275994
- [Background] Hanna N, Neubauer M, Yiannoutsos C, McGarry R, Arseneau J, Ansari R, Reynolds C, Govindan R, Melnyk A, Fisher W, Richards D, Bruetman D, Anderson T, Chowhan N, Nattam S, Mantravadi P, Johnson C, Breen T, White A, Einhorn L; Hoosier Oncology Group; US Oncology. Phase III study of cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel in patients with inoperable stage III non-small-cell lung cancer: the Hoosier Oncology Group and U.S. Oncology. J Clin Oncol. 2008 Dec 10;26(35):5755-60. doi: 10.1200/JCO.2008.17.7840. Epub 2008 Nov 10. PMID 19001323
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369